CLINICAL TRIAL: NCT05357859
Title: Effect of Vitamin D Supplement for Cognitive Function in Patients With Bipolar Disorder- Randomized Double-Blind Controlled Trial
Brief Title: Vitamin D for Cognition in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Wen Yin Chen, Psychiatrist in Taipei City Hospital, songde branch, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vitamin D in bipolar
Record Dates: First submitted 2022-04-18; First posted 2022-05-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; vitamin D; cognition
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: double blinded RCT
Who Masked: Participant, Care Provider
Masking Description: A pharmacist will prepare the dosing of solubilized vitamin D3 and also identical appearance of placebo according to a randomized block schedule. Patients and researchers were blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: solubilized vitamin D3 in MCT (Experimental): The intervention dose and duration aims to correct their vitamin D deficiency to sufficient status (total serum 25(OH)D >/=30 ng/mL or 75 nmol/L). According to an oral cholecalciferol (D3) loading dose guideline for vitamin D-deficient adults (van Groningen et al. 2010), cumulative dose of more than 200,000 IU solubilized vitamin D3 would be applied in current RCT, with make sure the sufficient supplement. Intervention group will receive 144,000 IU in week0 (W0) and then every 2 weeks of 72,000 IU for total 8 weeks (totally 5 times: 144,000 IU wk0/ 72,000 IU wk2/ 72,000 IU wk4/ 72,000 IU wk6/ 72,000 IU wk8), theoretically to achieve sufficient levels of vitamin D.
  Interventions: Dietary Supplement: solubilized vitamin D3
- Placebo: MCT with same amount (Placebo Comparator): control group will receive same volume amount of medium chain triglyceride (MCT).
  Interventions: Dietary Supplement: medium chain triglyceride

INTERVENTIONS:
Dietary Supplement: solubilized vitamin D3 — solubilized vitamin D3
  Arms: Intervention: solubilized vitamin D3 in MCT
Dietary Supplement: medium chain triglyceride — MCT with same amount
  Arms: Placebo: MCT with same amount

SUMMARY:
Conduct randomized double-blind controlled trial (RCT), to examine the effects of vitamin D on cognitive performance in euthymic BD.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic mental disease related to recurrent episodes along with cognitive or functional decline. Comparing efficacy of pharmacological interventions targeting to treat cognitive deficit in BD is unexplored. The majority of the observational studies demonstrate a significant association between low serum vitamin D and compromised cognition in a wide range of neuropsychiatry diseases. Recent survey further revealed the high prevalence of hypovitamin D in BD. The effect of supplement and association between vitamin D and cognition in BD and the underlying mechanism is unclear.

The investigators will collect vitamin D levels and assess their association with cognition in a euthymic bipolar cohort (N=200) for screen. Then, the investigators estimate to recruit 120 of participants with cognitive deficits and combined vitamin D deficiency, to conduct a RCT. Participants will keep their usual treatment and will be randomized to receive either vitamin D supplement or a placebo for eight weeks. Cognitive test, adverse side effect, mood status and blood 25(OH)D levels and biomarkers will be measured before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who diagnosed with BD-I based on the Diagnostic and Statistical Manual (DSM-IV) criteria are consecutively referred by board-certified psychiatrists in Taipei City Hospital, Songde branch.
2. Age of participants should range from 20 to 65 years old.
3. No history of vitamin D supplementation within three months before the study.
4. The BD patients in their euthymic state (both Hamilton Depression Rating Scale and Young Mania Rating Scale ≤ 8) and no change of their psychoactive medications in recent three months.

Exclusion Criteria:

1. With known substance use disorder (except nicotine use disorder)
2. With any disorder with known neurological symptoms or complications (ex. brain injury, stroke or brain lesions)
3. Comorbid with schizophrenia spectrum disorders
4. With active physical condition (such as renal impairment, hepatic failure…) or pregnancy
5. Inability to complete the standard assessment or incapability of providing informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
change of cognition | Week 0, Week 10
  Change from Baseline Brief Assessment of Cognition in Affective Disorders (BAC-A) score at week 10

SECONDARY OUTCOMES:
change of serum vitamin D levels | Week 0, Week 10
  change from baseline serum vitamin D levels to week 10, unit: ng/mL
change of serum creatinine | Week 0, Week 10
  change from baseline serum creatinine to week 10, unit: mg/dL
change of blood albumin | Week 0, Week 10
  change from baseline blood albumin to week 10, unit: g/dL
change of blood parathyroid hormone | Week 0, Week 10
  change from baseline parathyroid hormone to week 10, unit: pg/mL
change of serum calcium levels | Week 0, Week 10
  change from baseline serum calcium levels to week 10, unit: mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
individual patient data can be sharing with de-identification process after asking